CLINICAL TRIAL: NCT03757000
Title: A Phase I Study of YY-20394 Given Orally to Patients With Relapsed or Refractory B Cell Hematologic Malignancies
Brief Title: A Phase I Study of YY-20394 in Patients With B Cell Hematologic Malignancies
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai YingLi Pharmaceutical Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YY-20394-001
Record Dates: First submitted 2018-11-16; First posted 2018-11-28 (Actual); Last update posted 2018-12-10 (Actual); Status verified 2018-12

CONDITIONS: B-cell Lymphoma Recurrent; B-cell Chronic Lymphocytic Leukemia
Keywords: YY-20394; B-cell Lymphoma Recurrent
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell

STUDY DESIGN:
Intervention Model Description: dose escalation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- YY-20394 (Experimental): YY-20394 is a selective inhibitor of the delta isoform of phosphatidylinositol 3- kinase (PI3Kδ).
  YY-20394 for clinical use is presented as a sterile tablets at 20 mg, or 100 mg doses. The drug product is intended for oral administration.Preset cohorts of 3-6 subjects will be enrolled sequentially at doses of 20, 40, 80, 140, 200, 260 and 320 mg/day.
  Interventions: Drug: YY-20394

INTERVENTIONS:
Drug: YY-20394 — YY-20394 is a new type of PI3K-δ selective inhibitor which differs structurally from idelalisib and its analogs, showing high potency against PI3Kδ, but with markedly improved selectivity (>1,000-fold selectivity for PI3K-δ versus PI3Kγ). This higher selectivity for PI3Kδ may decrease the risk of serious infection seen with idelalisib and especially with duvelisib due to strong immune suppression.Preclinical evaluation has demonstrated improved efficacy and safety for YY-20394 compared to idelalisib.

SUMMARY:
Protocol YY-20394-001 is a phase I open-label, first in human, dose escalation study to assess the tolerability, pharmacokinetics (PK) and efficacy of YY-20394 in patients with relapse or refractory B cell malignant hematological tumor.

DETAILED DESCRIPTION:
This is a two-part study comprised of a dose escalation part and a dose expansion part.

In the dose escalation part single patient cohorts will be dosed until a single related toxicity of Grade ≥ 3 or a Dose Limiting Toxicity (DLT) is observed. If this occurs, the study will switch to a conventional oncology 3+3 design (3 patients per dose cohort, with the potential to add an additional 3 patients if toxicity is observed) and escalation will continue until the maximum tolerated dose (MTD) is reached and a recommended Phase II (RP2D) dose is determined. Once the MTD is established a separate dose expansion part will enroll up total additional 12 patients at the RP2D.

In this clinical trial, YY-20394 is given orally once daily. A treatment cycle is defined as 28 days. YY-20394 was given until disease progression, unacceptable toxicity, or withdrawal from the study. The protocol was initiated with a single-patient cohort, treated with oral YY-20394 20 mg once daily (QD). Subsequent cohorts used a 3+3 design and evaluated doses of 40-320mg QD. Adverse events (AEs) were graded by NCI-CTCAE v4.0. Efficacy was assessed according to IWG-NHL and CLL consensus response criteria.

ELIGIBILITY:
Inclusion Criteria:

1. Males and/or females over age 18
2. Histologically or cytologically confirmed B cell malignancies
3. Eastern Cooperative Oncology Group performance status of 0 to 2
4. Life expectancy of at least 3 months
5. At least one measurable lesion by Computed Tomography(CT) or Magnetic Resonance Imaging(MRI) according to, which is not in irradiated area (only for expansion phase)
6. Acceptable hematologic status:

   Absolute neutrophil count(ANC)≥1.0×109/L; Platelet count(PLT)≥70×109/L; Hemoglobin(Hb)≥80 g/L; Total bilirubin(TBIL)≤1.5×Upper limit of normal value(ULN); Alanine aminotransferase(ALT)≤1.5×ULN; Aspartate aminotransferase(AST)≤1.5×ULN; Blood urea nitrogen(BUN)≤1×ULN; Creatinine(Cr)≤1×ULN; Left Ventricular Ejection Fractions(LVEF)≥50%； QTcF：male<450 ms,female<470 ms
7. The washout period from the last time accepting any anti-tumor treatment (including radiation therapy, chemotherapy, hormone therapy, surgery, or molecular targeted therapy) to participating in this test should be 4 weeks or more.
8. The last time participate in an investigational drug or device study should be more than one month prior to study entry.
9. Ability to understand the purposes and risks of the study
10. Availability of the signed informed consent forms (ICFs) approved by the investigator's Institutional Review Board (IRB)/Independent Ethics Committee (IEC) of the study site obtained before entering the study.

Exclusion Criteria:

1. Previously treated with PI3Kδ inhibitors and cause disease progression.
2. Any anti-tumor treatment, within 4 weeks prior to study entry.
3. There are third interstitial effusions (such as massive pleural effusion and ascites) which can not be controlled by drainage or other methods.
4. The dosage of steroid hormone (prednisone equivalent) was greater than 20mg/ days, and lasted for more than 14 days.
5. Medical history of difficulty in swallowing, malabsorption, or other chronic gastrointestinal disease, or conditions that may hamper compliance and/or absorption of the tested product.
6. During the study period, drugs that may prolong the QT (such as anti arrhythmic drugs) could not be interrupted.
7. Patients with central nervous system (CNS) involvement.
8. Allergy, or known to be allergic to the drug.
9. Active, uncontrolled bacterial, viral, or fungal infections, requiring systemic therapy(such as pneumonia).
10. Known infection with human immunodeficiency virus (HIV), hepatitis B virus(HBV), or hepatitis C virus (HCV).
11. History of immunodeficiency, including HIV positive test, other acquired or congenital immunodeficiency disorders, organ transplantation or allogeneic bone marrow transplantation.
12. Autologous hematopoietic stem cell transplantation was received within 90 days before the first dose treatment.
13. Has suffered from any heart disease, including: (1) angina pectoris; (2) medicated or clinically significant arrhythmia; (3) myocardial infarction; (4) heart failure; (5) any other heart disease judged by the researchers not suitable for the test.
14. The baseline pregnancy test was positive in pregnant women, lactating women or fertile women.
15. According to the judgement of the researcher, there are concomitant diseases that seriously endanger the safety of patients or affect the completion of the study (such as severe hypertension, diabetes, thyroid diseases, etc.).
16. Receiving granulocyte colony-stimulating factor(GCSF) or blood transfusion within 7 days before screening.
17. Patients suffering from other primary malignant tumors in the past 5 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2017-12-25 (Actual); Primary Completion 2019-03-30 (Estimated); Study Completion 2019-05-30 (Estimated)

PRIMARY OUTCOMES:
Dose limited toxicities evaluated with NCI-CTC AE v4.0 | within 28 days after the first dose
  Incidence of dose limited toxicities and associated dose of YY-20394
Adverse events evaluated by NCI CTCAE v4.0 | from the first dose to within 30 days after the last dose
  Incidence of adverse events and associated dose of YY-20394

SECONDARY OUTCOMES:
Plasma concentration of YY-20394 | within 56 days after the first dose
  This composite endpoint will measure the plasma concentration of YY-20394.
Objective response rate | within 30 days after the last dose
  the proportion of subjects who have a Complete Response or Partial Response
Disease control rate | within 30 days after the last dose
  the proportion of subjects who have a Complete Response or Partial Response

CONTACTS AND LOCATIONS:
Overall Officials: Hanying Bao, PhD, Study Director — Shanghai YingLi Pharmaceutical Co. Ltd.
Locations (3):
- China (3):
  - Peking Cancer Hospital, Beijing, Beijing Municipality
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - Hematology Hospital of Chinese Academy of Medical Sciences, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Eisenreich A, Rauch U. PI3K inhibitors in cardiovascular disease. Cardiovasc Ther. 2011 Feb;29(1):29-36. doi: 10.1111/j.1755-5922.2010.00206.x. PMID 20626398
- [Result] Samuels Y, Wang Z, Bardelli A, Silliman N, Ptak J, Szabo S, Yan H, Gazdar A, Powell SM, Riggins GJ, Willson JK, Markowitz S, Kinzler KW, Vogelstein B, Velculescu VE. High frequency of mutations of the PIK3CA gene in human cancers. Science. 2004 Apr 23;304(5670):554. doi: 10.1126/science.1096502. Epub 2004 Mar 11. No abstract available. PMID 15016963
- [Result] Yuan TL, Cantley LC. PI3K pathway alterations in cancer: variations on a theme. Oncogene. 2008 Sep 18;27(41):5497-510. doi: 10.1038/onc.2008.245. PMID 18794884
- [Result] Kong D, Yamori T. Phosphatidylinositol 3-kinase inhibitors: promising drug candidates for cancer therapy. Cancer Sci. 2008 Sep;99(9):1734-40. doi: 10.1111/j.1349-7006.2008.00891.x. Epub 2008 Jul 4. PMID 18616528
- [Result] Brown JR, Byrd JC, Coutre SE, Benson DM, Flinn IW, Wagner-Johnston ND, Spurgeon SE, Kahl BS, Bello C, Webb HK, Johnson DM, Peterman S, Li D, Jahn TM, Lannutti BJ, Ulrich RG, Yu AS, Miller LL, Furman RR. Idelalisib, an inhibitor of phosphatidylinositol 3-kinase p110delta, for relapsed/refractory chronic lymphocytic leukemia. Blood. 2014 May 29;123(22):3390-7. doi: 10.1182/blood-2013-11-535047. Epub 2014 Mar 10. PMID 24615777
- [Result] Flinn IW, Kahl BS, Leonard JP, Furman RR, Brown JR, Byrd JC, Wagner-Johnston ND, Coutre SE, Benson DM, Peterman S, Cho Y, Webb HK, Johnson DM, Yu AS, Ulrich RG, Godfrey WR, Miller LL, Spurgeon SE. Idelalisib, a selective inhibitor of phosphatidylinositol 3-kinase-delta, as therapy for previously treated indolent non-Hodgkin lymphoma. Blood. 2014 May 29;123(22):3406-13. doi: 10.1182/blood-2013-11-538546. Epub 2014 Mar 10. PMID 24615776
- [Result] Gopal AK, Kahl BS, de Vos S, Wagner-Johnston ND, Schuster SJ, Jurczak WJ, Flinn IW, Flowers CR, Martin P, Viardot A, Blum KA, Goy AH, Davies AJ, Zinzani PL, Dreyling M, Johnson D, Miller LL, Holes L, Li D, Dansey RD, Godfrey WR, Salles GA. PI3Kdelta inhibition by idelalisib in patients with relapsed indolent lymphoma. N Engl J Med. 2014 Mar 13;370(11):1008-18. doi: 10.1056/NEJMoa1314583. Epub 2014 Jan 22. PMID 24450858
- [Result] Furman RR, Sharman JP, Coutre SE, Cheson BD, Pagel JM, Hillmen P, Barrientos JC, Zelenetz AD, Kipps TJ, Flinn I, Ghia P, Eradat H, Ervin T, Lamanna N, Coiffier B, Pettitt AR, Ma S, Stilgenbauer S, Cramer P, Aiello M, Johnson DM, Miller LL, Li D, Jahn TM, Dansey RD, Hallek M, O'Brien SM. Idelalisib and rituximab in relapsed chronic lymphocytic leukemia. N Engl J Med. 2014 Mar 13;370(11):997-1007. doi: 10.1056/NEJMoa1315226. Epub 2014 Jan 22. PMID 24450857
- [Derived] Jiang B, Qi J, Song Y, Li Z, Tu M, Ping L, Liu Z, Bao H, Xu Z, Qiu L. Phase 1 clinical trial of the PI3Kdelta inhibitor YY-20394 in patients with B-cell hematological malignancies. J Hematol Oncol. 2021 Aug 23;14(1):130. doi: 10.1186/s13045-021-01140-z. PMID 34425850
- See also: Related Info — http://www.wanfangdata.com.cn/details/detail.do?_type=conference&id=7408347
- See also: Related Info — http://www.wanfangdata.com.cn/details/detail.do?_type=perio&id=ez200803022